CLINICAL TRIAL: NCT03065556
Title: A Double-Blind, Randomized, Multicenter, Vehicle-Controlled, Parallel Group Study to Determine the Efficacy and Safety of 188-0551 in Subjects With Plaque Psoriasis Receiving Up To Four Weeks of Twice-Daily Treatment
Brief Title: A Comparison of 188-0551 Solution Versus Vehicle Solution in Subjects With Plaque Psoriasis (Study 203)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 188-0551-203
Record Dates: First submitted 2017-02-16; First posted 2017-02-28 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 188-0551 Solution (Experimental): 188-0551 Solution applied topically twice daily
  Interventions: Drug: 188-0551 Solution
- Vehicle Solution (Placebo Comparator): Vehicle Solution applied topically twice daily
  Interventions: Drug: Vehicle Solution

INTERVENTIONS:
Drug: 188-0551 Solution — Topical solution containing active drug
  Arms: 188-0551 Solution
Drug: Vehicle Solution — Topical solution containing no active drug
  Arms: Vehicle Solution

SUMMARY:
This Phase 2 study (Study 203) has been designed to determine and compare the efficacy and safety of 188-0551 Solution and Vehicle Solution applied twice daily for up to four weeks in subjects with plaque psoriasis. Subjects will be instructed to apply the test article (188-0551 Solution or Vehicle Solution) to all psoriasis plaques within the designated Treatment Area twice daily for four weeks (Study Day 29), unless the investigator verifies the subject's psoriasis has cleared at Day 15, then test article application will be for 2 weeks (Study Day 15).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or non-pregnant female and is at least 18 years of age.
2. Subject has provided written informed consent.
3. Subject is willing and able to apply the test article(s) as directed.
4. Subject has a clinical diagnosis of stable plaque psoriasis.
5. Subject has an Investigator's Global Assessment (IGA) score of at least three (3 = moderate) at the Baseline Visit.
6. Females must be post-menopausal, surgically sterile or use an effective method of birth control, with a negative urine pregnancy test (UPT) at the Baseline Visit.

Exclusion Criteria:

1. Subject has spontaneously improving or rapidly deteriorating plaque psoriasis.
2. Subject has guttate, pustular, erythrodermic or other non-plaque forms of psoriasis.
3. Subject has a physical condition which, in the investigator's opinion, might impair evaluation of plaque psoriasis.
4. Subject has used any phototherapy (including laser), photo-chemotherapy or other forms of photo based therapy for the treatment of their psoriasis within 30 days prior to the Baseline Visit.
5. Subject has used any systemic tofacitinib, apremilast, methotrexate, retinoids, systemic corticosteroids [including intralesional, intra-articular, and intramuscular corticosteroids], cyclosporine or analogous products within 90 days prior to the Baseline Visit.
6. Subject has used any systemic anti-inflammatory biologic therapy.
7. Subject had prolonged exposure to natural or artificial sources of ultraviolet radiation within 30 days prior to the Baseline Visit or is intending to have such exposure during the study which in the opinion of the investigator is thought to modify the subject's disease.
8. Subject has used topical body (excluding the scalp) psoriasis therapy (including coal tar, anthralin, steroids, retinoids and vitamin D analogs) within 14 days prior to the Baseline Visit.
9. Subject has used emollients/moisturizers on areas to be treated within four hours prior to clinical evaluation at the Baseline Visit.
10. Subject is currently using lithium or Plaquenil (hydroxychloroquine).
11. Subject is currently using a beta-blocking medication (e.g., propranolol) or angiotensin converting enzyme (ACE) inhibitor at a dose that has not been stabilized, in the opinion of the investigator.
12. Subject has a history of sensitivity to corticosteroids or any of the ingredients in the test articles.
13. Subject is pregnant, lactating, or is planning to become pregnant during the study.
14. Subject is currently enrolled in an investigational drug or device study.
15. Subject has used an investigational drug or investigational device treatment within 30 days prior to the Baseline Visit.
16. Subject has been previously enrolled in this study and treated with a test article.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects rated a treatment success based on the Investigator's Global Assessment (IGA) | End of Study (Day 15 or 29)
  The primary efficacy endpoint will be the proportion of subjects with IGA treatment success at EOS where EOS is the subject's last completed post-Baseline visit (Day 15 or 29).

SECONDARY OUTCOMES:
Proportion of subjects rated a treatment success for each of the clinical signs of psoriasis (scaling, erythema and plaque elevation) | End of Study (Day 15 or 29)
  Scaling, erythema and plaque elevation will each be scored on a 5-point scale where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe. These evaluations are an assessment of the overall or "average" degree of each of three key characteristics present within all of the subject's psoriatic lesions in the Treatment Area by the investigator or designee.
Change from Baseline in pruritus score | End of Study (Day 15 or 29)
  At the Baseline Visit, prior to the first application of the test article, the subject's overall experience of pruritus within the previous two (2) weeks will be assessed using a questionnaire that assesses the degree, duration, direction, disability, and distribution of the subject's pruritus. At Days 15 and 29, the overall experience of pruritus, in the previous two weeks, will be scored using the same questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Site 01, Arlington Heights, Illinois, United States

IPD SHARING:
Plan to Share IPD: No